CLINICAL TRIAL: NCT03960645
Title: A Phase 1b, Open-label Study to Evaluate the PK, Safety and Efficacy of B/F/TAF in HIV-1 Infected, Virologically Suppressed, Pregnant Women in Their Second and Third Trimesters
Brief Title: Study to Evaluate the Pharmacokinetics (PK), Safety, and Efficacy of B/F/TAF in Human Immunodeficiency Virus (HIV)-1 Infected, Virologically Suppressed, Pregnant Women in Their Second and Third Trimesters
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-380-5310; 2021-001073-23 (EudraCT Number)
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2023-12

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: Study model 'single group' is selected as the Neonates group was only followed up but not treated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- B/F/TAF (Experimental): Pregnant women participants will receive fixed dose combination (FDC) tablet of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) 50/200/25 mg for up to 38 weeks (from the second or third trimesters of pregnancy, depending on enrollment, through 12 weeks post-partum).
  Interventions: Drug: B/F/TAF
- Neonates (No Intervention): Neonates who will be born to women participants in the study will be followed from birth up to 8 weeks of age after obtaining consent from the parent or legal guardian. None of the neonates that participate in the study will be treated with the study drug.

INTERVENTIONS:
Drug: B/F/TAF — 50/200/25 mg FDC tablet administered orally once daily without regard to food.
  Other Names: GS-9883/F/TAF, Biktarvy®, BVY
  Arms: B/F/TAF

SUMMARY:
The primary objective of this study is to evaluate the steady state PK of bictegravir (BIC) and confirm the dose of BIC/emtricitabine/tenofovir alafenamide (B/F/TAF) 50/200/25 mg fixed dose combination (FDC) in HIV-1 infected, virologically suppressed pregnant women in their second and third trimesters.

ELIGIBILITY:
Key Inclusion Criteria:

* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures
* With singleton pregnancy, at least 12 weeks but not more than 31 weeks pregnant at the time of screening
* Agree not to breastfeed for the duration of the study
* Currently on a stable antiretroviral regimen for ≥ 6 months preceding the screening visit
* Documented plasma HIV-1 ribonucleic acid (RNA) levels of < 50 copies/mL for ≥ 6 months preceding the screening visit and have HIV-1 RNA < 50 copies/mL at the screening visit
* Have no documented or suspected resistance to FTC, Tenofovir (TFV), or integrase strand-transfer inhibitors (INSTIs) including, but not limited to, the reverse transcriptase resistance mutations K65R or M184V/I
* Have a normal ultrasound, completed locally prior to the Day 1 visit, with no evidence of any fetal malformation or structural abnormality affecting either fetus or placenta
* Normal maternal alfa-fetoprotein level at the screening visit

Key Exclusion Criteria:

* Have chronic hepatitis B virus (HBV)
* Have active hepatitis C virus (HCV) infection
* An opportunistic illness indicative of stage 3 HIV diagnosed within the 30 days prior to screening

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 62 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (8):
- United States (2):
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
- Instituto Dominicano de Estudios Virologics (IDEV), Santo Domingo, Dominican Republic
- Thailand (5):
  - Faculty of Medicine Siriraj Hospital, Bangkok Noi
  - Faculty of Medicine-Khon Kaen University, Khon Kaen
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi
  - Research Institute for Health Sciences, Chiang Mai University, Nonthaburi
  - Thai Red Cross AIDS Research Centre, Pathumwan

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gileadclinicaltrials.com/transparency-policy#Commitment
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gileadclinicaltrials.com/transparency-policy#Commitment

REFERENCES:
- [Derived] Zhang H, Hindman JT, Lin L, Davis M, Shang J, Xiao D, Avihingsanon A, Arora P, Palaparthy R, Girish S, Marathe DD. A study of the pharmacokinetics, safety, and efficacy of bictegravir/emtricitabine/tenofovir alafenamide in virologically suppressed pregnant women with HIV. AIDS. 2024 Jan 1;38(1):F1-F9. doi: 10.1097/QAD.0000000000003783. Epub 2023 Nov 22. PMID 37939141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the Dominican Republic, Thailand and the United States.
Pre-assignment Details: 33 pregnant women were enrolled in the B/F/TAF group. Neonates born to these women were also enrolled in the study for follow up. A total of 29 neonate participants were enrolled.
Groups:
- B/F/TAF: Pregnant women participants received fixed dose combination (FDC) tablet of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) 50/200/25 mg, orally, once daily for up to 38 weeks (from the second or third trimesters of pregnancy, depending on enrollment, through 12 weeks post-partum).
- Neonates: Neonates born to women participants in the study were followed from birth up to 8 weeks of age after obtaining consent from the parent or legal guardian. None of the neonates participating in the study were treated with the study drug.
Period: Overall Study
Arm/Group | B/F/TAF | Neonates
Started | 33 | 29
Completed | 32 | 29
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: B/F/TAF: Safety analysis set included all adult participants who took at least 1 dose of study drug (B/F/TAF). Neonates: Safety analysis set included neonates who were born to women participating in the study and had been enrolled into the study as well.
Groups:
- B/F/TAF: Pregnant women participants received FDC tablet of B/F/TAF 50/200/25 mg, orally, once daily for up to 38 weeks (from the second or third trimesters of pregnancy, depending on enrollment, through 12 weeks post-partum).
- Total: Total of all reporting groups
Arm/Group | B/F/TAF | Neonates | Total
Number analyzed (Participants) | 33 | 29 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (5.0) | 0 (0.0) | 16 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 10 | 43
  Male | 0 | 19 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 29 | 25 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 25 | 24 | 49
  Race: Black | 6 | 4 | 10
  Race: Other | 1 | 1 | 2
  Race: White | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Thailand | 25 | 24 | 49
  United States | 5 | 2 | 7
  Dominican Republic | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of Bictegravir (BIC)
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: Intensive PK: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours postdose in second trimester (Weeks 20-28), third trimester (Weeks 30-38), Week 6 post-partum, and Week 12 post-partum
Population: PK analysis set included all enrolled adult participants who took at least 1 dose of study drug (B/F/TAF), and had at least 1 non-missing concentration value reported by the PK laboratory for the corresponding analytes (BIC, FTC, TAF, and tenofovir diphosphate [TFV-DP]). Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
hours*nanograms per milliliter (h*ng/mL)
  Second Trimester: number analyzed (Participants) | 20
  Second Trimester | 62772.2 (20242.18)
  Third Trimester: number analyzed (Participants) | 30
  Third Trimester | 60163.4 (17482.06)
  Week 6 Post-partum: number analyzed (Participants) | 31
  Week 6 Post-partum | 134820.3 (36217.30)
  Week 12 Post-partum | 148251.6 (42189.17)
Statistical Analysis 1: Comparison: B/F/TAF; BIC: Second Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% confidence interval (CI) was constructed for the geometric least squares mean (GLSM) ratio (%); Test type: Other; GLSM ratio (%) = 41.24, 90% CI 2-sided [36.71 to 46.32]
Statistical Analysis 2: Comparison: B/F/TAF; BIC: Second Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 44.65, 90% CI 2-sided [40.04 to 49.79]
Statistical Analysis 3: Comparison: B/F/TAF; BIC: Third Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 40.57, 90% CI 2-sided [36.77 to 44.76]
Statistical Analysis 4: Comparison: B/F/TAF; BIC: Third Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 44.40, 90% CI 2-sided [39.95 to 49.34]

2. Secondary Outcome: PK Parameter: AUCtau of Emtricitabine (FTC) and Tenofovir Alafenamide (TAF)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
h*ng/mL
  FTC: Second Trimester: number analyzed (Participants) | 21
  FTC: Second Trimester | 10263.8 (2054.35)
  FTC: Third Trimester: number analyzed (Participants) | 30
  FTC: Third Trimester | 10435.2 (2121.87)
  FTC: Week 6 Post-partum: number analyzed (Participants) | 31
  FTC: Week 6 Post-partum | 16277.5 (4023.42)
  FTC: Week 12 Post-partum | 15308.5 (3359.83)
  TAF: Second Trimester: number analyzed (Participants) | 15
  TAF: Second Trimester | 235.5 (107.36)
  TAF: Third Trimester: number analyzed (Participants) | 17
  TAF: Third Trimester | 212.1 (95.38)
  TAF: Week 6 Post-partum: number analyzed (Participants) | 27
  TAF: Week 6 Post-partum | 374.3 (153.54)
  TAF: Week 12 Post-partum: number analyzed (Participants) | 30
  TAF: Week 12 Post-partum | 296.4 (94.37)
Statistical Analysis 1: Comparison: B/F/TAF; FTC: Second Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 67.38, 90% CI 2-sided [63.45 to 71.56]
Statistical Analysis 2: Comparison: B/F/TAF; FTC: Second Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 64.26, 90% CI 2-sided [60.95 to 67.75]
Statistical Analysis 3: Comparison: B/F/TAF; FTC: Third Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 69.19, 90% CI 2-sided [65.88 to 72.66]
Statistical Analysis 4: Comparison: B/F/TAF; FTC: Third Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 65.09, 90% CI 2-sided [61.79 to 68.57]
Statistical Analysis 5: Comparison: B/F/TAF; TAF: Second Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 77.62, 90% CI 2-sided [65.40 to 92.14]
Statistical Analysis 6: Comparison: B/F/TAF; TAF: Second Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 62.50, 90% CI 2-sided [50.76 to 76.96]
Statistical Analysis 7: Comparison: B/F/TAF; TAF: Third Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 69.67, 90% CI 2-sided [58.57 to 82.88]
Statistical Analysis 8: Comparison: B/F/TAF; TAF: Third Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 56.52, 90% CI 2-sided [46.32 to 68.96]

3. Secondary Outcome: PK Parameter: AUClast of BIC, FTC, and TAF
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: as for outcome 1
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
h*ng/mL
  BIC: Second Trimester: number analyzed (Participants) | 21
  BIC: Second Trimester | 63187.5 (19814.99)
  BIC: Third Trimester: number analyzed (Participants) | 30
  BIC: Third Trimester | 60145.3 (17484.52)
  BIC: Week 6 Post-partum: number analyzed (Participants) | 31
  BIC: Week 6 Post-partum | 135058.9 (36348.21)
  BIC: Week 12 Post-partum | 148265.3 (42201.47)
  FTC: Second Trimester: number analyzed (Participants) | 21
  FTC: Second Trimester | 10258.5 (2049.53)
  FTC: Third Trimester: number analyzed (Participants) | 30
  FTC: Third Trimester | 10434.2 (2121.13)
  FTC: Week 6 Post-partum: number analyzed (Participants) | 31
  FTC: Week 6 Post-partum | 16329.7 (4095.44)
  FTC: Week 12 Post-partum | 15308.5 (3359.79)
  TAF: Second Trimester: number analyzed (Participants) | 21
  TAF: Second Trimester | 220.4 (98.98)
  TAF: Third Trimester: number analyzed (Participants) | 30
  TAF: Third Trimester | 202.2 (84.98)
  TAF: Week 6 Post-partum: number analyzed (Participants) | 31
  TAF: Week 6 Post-partum | 356.7 (151.27)
  TAF: Week 12 Post-partum | 294.3 (97.88)

4. Secondary Outcome: PK Parameter: Cmax of BIC, FTC, and TAF
Description: Cmax is defined as the maximum observed concentration of drug during the dosing interval.
Time Frame: as for outcome 1
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
ng/mL
  BIC: Second Trimester: number analyzed (Participants) | 21
  BIC: Second Trimester | 5819.0 (1752.29)
  BIC: Third Trimester: number analyzed (Participants) | 30
  BIC: Third Trimester | 5374.7 (1393.86)
  BIC: Week 6 Post-partum: number analyzed (Participants) | 31
  BIC: Week 6 Post-partum | 9765.5 (2274.93)
  BIC: Week 12 Post-partum | 11025.3 (2747.42)
  FTC: Second Trimester: number analyzed (Participants) | 21
  FTC: Second Trimester | 2639.1 (965.60)
  FTC: Third Trimester: number analyzed (Participants) | 30
  FTC: Third Trimester | 2586.0 (686.42)
  FTC: Week 6 Post-partum: number analyzed (Participants) | 31
  FTC: Week 6 Post-partum | 3394.8 (951.83)
  FTC: Week 12 Post-partum | 3360.0 (902.47)
  TAF: Second Trimester: number analyzed (Participants) | 21
  TAF: Second Trimester | 332.4 (173.29)
  TAF: Third Trimester: number analyzed (Participants) | 30
  TAF: Third Trimester | 270.9 (113.93)
  TAF: Week 6 Post-partum: number analyzed (Participants) | 31
  TAF: Week 6 Post-partum | 506.4 (249.33)
  TAF: Week 12 Post-partum | 494.6 (259.51)
Statistical Analysis 1: Comparison: B/F/TAF; BIC: Second Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 51.91, 90% CI 2-sided [46.48 to 57.97]
Statistical Analysis 2: Comparison: B/F/TAF; BIC: Second Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 57.67, 90% CI 2-sided [52.48 to 63.36]
Statistical Analysis 3: Comparison: B/F/TAF; BIC: Third Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 48.18, 90% CI 2-sided [43.03 to 53.94]
Statistical Analysis 4: Comparison: B/F/TAF; BIC: Third Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 54.42, 90% CI 2-sided [48.39 to 61.21]
Statistical Analysis 5: Comparison: B/F/TAF; FTC: Second Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 75.61, 90% CI 2-sided [66.70 to 85.70]
Statistical Analysis 6: Comparison: B/F/TAF; FTC: Second Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 77.81, 90% CI 2-sided [68.76 to 88.05]
Statistical Analysis 7: Comparison: B/F/TAF; FTC: Third Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 77.45, 90% CI 2-sided [70.33 to 85.29]
Statistical Analysis 8: Comparison: B/F/TAF; FTC: Third Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 77.08, 90% CI 2-sided [69.78 to 85.15]
Statistical Analysis 9: Comparison: B/F/TAF; TAF: Second Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 69.90, 90% CI 2-sided [56.16 to 87.00]
Statistical Analysis 10: Comparison: B/F/TAF; TAF: Second Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 66.55, 90% CI 2-sided [53.79 to 82.34]
Statistical Analysis 11: Comparison: B/F/TAF; TAF: Third Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 57.14, 90% CI 2-sided [46.04 to 70.91]
Statistical Analysis 12: Comparison: B/F/TAF; TAF: Third Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 55.27, 90% CI 2-sided [44.65 to 68.42]

5. Secondary Outcome: PK Parameter: Ctau of BIC and FTC
Description: Ctau is defined as the observed drug concentration at the end of the dosing interval.
Time Frame: as for outcome 1
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
ng/mL
  BIC: Second Trimester: number analyzed (Participants) | 20
  BIC: Second Trimester | 1046.4 (472.68)
  BIC: Third Trimester: number analyzed (Participants) | 30
  BIC: Third Trimester | 1072.4 (447.03)
  BIC: Week 6 Post-partum: number analyzed (Participants) | 31
  BIC: Week 6 Post-partum | 3530.3 (1354.20)
  BIC: Week 12 Post-partum | 3641.9 (1241.64)
  FTC: Second Trimester: number analyzed (Participants) | 21
  FTC: Second Trimester | 59.8 (62.17)
  FTC: Third Trimester: number analyzed (Participants) | 30
  FTC: Third Trimester | 51.4 (13.98)
  FTC: Week 6 Post-partum: number analyzed (Participants) | 31
  FTC: Week 6 Post-partum | 152.1 (271.50)
  FTC: Week 12 Post-partum | 81.1 (27.34)
Statistical Analysis 1: Comparison: B/F/TAF; BIC: Second Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 26.17, 90% CI 2-sided [21.45 to 31.93]
Statistical Analysis 2: Comparison: B/F/TAF; BIC: Second Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 26.99, 90% CI 2-sided [22.23 to 32.78]
Statistical Analysis 3: Comparison: B/F/TAF; BIC: Third Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 29.03, 90% CI 2-sided [25.74 to 32.74]
Statistical Analysis 4: Comparison: B/F/TAF; BIC: Third Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 29.97, 90% CI 2-sided [26.47 to 33.93]
Statistical Analysis 5: Comparison: B/F/TAF; FTC: Second Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 64.22, 90% CI 2-sided [54.63 to 75.49]
Statistical Analysis 6: Comparison: B/F/TAF; FTC: Second Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 42.89, 90% CI 2-sided [36.55 to 50.34]
Statistical Analysis 7: Comparison: B/F/TAF; FTC: Third Trimester (Test) vs. Week 12 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 64.71, 90% CI 2-sided [59.30 to 70.61]
Statistical Analysis 8: Comparison: B/F/TAF; FTC: Third Trimester (Test) vs. Week 6 Post-partum (Reference). A 90% CI was constructed for the GLSM ratio (%); Test type: Other; GLSM ratio (%) = 46.92, 90% CI 2-sided [39.57 to 55.64]

6. Secondary Outcome: PK Parameter: Clast of BIC, FTC, and TAF
Description: Clast is defined as the last observable concentration of drug.
Time Frame: as for outcome 1
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
ng/mL
  BIC: Second Trimester: number analyzed (Participants) | 21
  BIC: Second Trimester | 1141.10 (631.431)
  BIC: Third Trimester: number analyzed (Participants) | 30
  BIC: Third Trimester | 1075.13 (447.847)
  BIC: Week 6 Post-partum: number analyzed (Participants) | 31
  BIC: Week 6 Post-partum | 3535.48 (1371.162)
  BIC: Week 12 Post-partum | 3641.88 (1240.605)
  FTC: Second Trimester: number analyzed (Participants) | 21
  FTC: Second Trimester | 75.08 (130.792)
  FTC: Third Trimester: number analyzed (Participants) | 30
  FTC: Third Trimester | 51.65 (14.182)
  FTC: Week 6 Post-partum: number analyzed (Participants) | 31
  FTC: Week 6 Post-partum | 156.16 (292.579)
  FTC: Week 12 Post-partum | 81.18 (27.334)
  TAF: Second Trimester: number analyzed (Participants) | 21
  TAF: Second Trimester | 4.49 (5.130)
  TAF: Third Trimester: number analyzed (Participants) | 30
  TAF: Third Trimester | 4.80 (4.048)
  TAF: Week 6 Post-partum: number analyzed (Participants) | 31
  TAF: Week 6 Post-partum | 3.13 (1.849)
  TAF: Week 12 Post-partum | 3.36 (1.999)

7. Secondary Outcome: PK Parameter: Tmax of BIC, FTC, and TAF
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: as for outcome 1
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
h
  BIC: Second Trimester: number analyzed (Participants) | 21
  BIC: Second Trimester | 2.00 [1.00 to 12.00]
  BIC: Third Trimester: number analyzed (Participants) | 30
  BIC: Third Trimester | 2.00 [1.00 to 6.00]
  BIC: Week 6 Post-partum: number analyzed (Participants) | 31
  BIC: Week 6 Post-partum | 1.50 [0.50 to 12.00]
  BIC: Week 12 Post-partum | 1.50 [0.50 to 4.00]
  FTC: Second Trimester: number analyzed (Participants) | 21
  FTC: Second Trimester | 1.50 [0.50 to 4.00]
  FTC: Third Trimester: number analyzed (Participants) | 30
  FTC: Third Trimester | 1.50 [0.50 to 4.00]
  FTC: Week 6 Post-partum: number analyzed (Participants) | 31
  FTC: Week 6 Post-partum | 1.50 [0.50 to 4.00]
  FTC: Week 12 Post-partum | 1.00 [0.50 to 3.00]
  TAF: Second Trimester: number analyzed (Participants) | 21
  TAF: Second Trimester | 0.75 [0.25 to 4.00]
  TAF: Third Trimester: number analyzed (Participants) | 30
  TAF: Third Trimester | 1.00 [0.25 to 3.00]
  TAF: Week 6 Post-partum: number analyzed (Participants) | 31
  TAF: Week 6 Post-partum | 0.75 [0.25 to 3.00]
  TAF: Week 12 Post-partum | 0.75 [0.25 to 3.00]

8. Secondary Outcome: PK Parameter: t1/2 of BIC, FTC, and TAF
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug.
Time Frame: as for outcome 1
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Median (Full Range); unit: h
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
h
  BIC: Second Trimester: number analyzed (Participants) | 19
  BIC: Second Trimester | 9.09 [4.75 to 16.04]
  BIC: Third Trimester: number analyzed (Participants) | 30
  BIC: Third Trimester | 9.91 [7.53 to 16.24]
  BIC: Week 6 Post-partum: number analyzed (Participants) | 29
  BIC: Week 6 Post-partum | 18.24 [12.18 to 29.59]
  BIC: Week 12 Post-partum: number analyzed (Participants) | 30
  BIC: Week 12 Post-partum | 17.27 [4.534 to 26.3]
  FTC: Second Trimester: number analyzed (Participants) | 20
  FTC: Second Trimester | 6.43 [4.76 to 7.36]
  FTC: Third Trimester: number analyzed (Participants) | 30
  FTC: Third Trimester | 6.41 [4.49 to 7.91]
  FTC: Week 6 Post-partum: number analyzed (Participants) | 28
  FTC: Week 6 Post-partum | 6.27 [4.47 to 7.80]
  FTC: Week 12 Post-partum | 5.76 [3.83 to 8.19]
  TAF: Second Trimester: number analyzed (Participants) | 14
  TAF: Second Trimester | 0.30 [0.22 to 0.66]
  TAF: Third Trimester: number analyzed (Participants) | 16
  TAF: Third Trimester | 0.28 [0.19 to 0.62]
  TAF: Week 6 Post-partum: number analyzed (Participants) | 26
  TAF: Week 6 Post-partum | 0.40 [0.25 to 0.60]
  TAF: Week 12 Post-partum: number analyzed (Participants) | 30
  TAF: Week 12 Post-partum | 0.35 [0.25 to 0.60]

9. Secondary Outcome: PK Parameter: CLss/F of BIC, FTC, and TAF
Description: CLss/F is defined as the apparent steady-state oral clearance following administration of the drug.
Time Frame: as for outcome 1
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
mL/h
  BIC: Second Trimester: number analyzed (Participants) | 20
  BIC: Second Trimester | 911.78 (433.301)
  BIC: Third Trimester: number analyzed (Participants) | 30
  BIC: Third Trimester | 902.47 (287.285)
  BIC: Week 6 Post-partum: number analyzed (Participants) | 31
  BIC: Week 6 Post-partum | 399.02 (113.214)
  BIC: Week 12 Post-partum | 362.40 (95.856)
  FTC: Second Trimester: number analyzed (Participants) | 21
  FTC: Second Trimester | 20228.02 (3981.186)
  FTC: Third Trimester: number analyzed (Participants) | 30
  FTC: Third Trimester | 19975.85 (4223.365)
  FTC: Week 6 Post-partum: number analyzed (Participants) | 31
  FTC: Week 6 Post-partum | 12991.62 (3111.349)
  FTC: Week 12 Post-partum | 13645.71 (2830.897)
  TAF: Second Trimester: number analyzed (Participants) | 15
  TAF: Second Trimester | 122677.74 (44270.041)
  TAF: Third Trimester: number analyzed (Participants) | 17
  TAF: Third Trimester | 135061.19 (44876.970)
  TAF: Week 6 Post-partum: number analyzed (Participants) | 27
  TAF: Week 6 Post-partum | 76939.32 (29189.555)
  TAF: Week 12 Post-partum: number analyzed (Participants) | 30
  TAF: Week 12 Post-partum | 92888.59 (29461.550)

10. Secondary Outcome: PK Parameter: Vz/F of BIC, FTC, and TAF
Description: Vz/F is defined as the apparent volume of distribution of the drug.
Time Frame: as for outcome 1
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
mL
  BIC: Second Trimester: number analyzed (Participants) | 19
  BIC: Second Trimester | 11896.24 (4417.149)
  BIC: Third Trimester: number analyzed (Participants) | 30
  BIC: Third Trimester | 13406.77 (4349.429)
  BIC: Week 6 Post-partum: number analyzed (Participants) | 29
  BIC: Week 6 Post-partum | 10348.47 (3713.380)
  BIC: Week 12 Post-partum: number analyzed (Participants) | 30
  BIC: Week 12 Post-partum | 8692.59 (2398.645)
  FTC: Second Trimester: number analyzed (Participants) | 20
  FTC: Second Trimester | 181767.32 (36739.344)
  FTC: Third Trimester: number analyzed (Participants) | 30
  FTC: Third Trimester | 184791.79 (56340.526)
  FTC: Week 6 Post-partum: number analyzed (Participants) | 28
  FTC: Week 6 Post-partum | 117384.90 (35385.941)
  FTC: Week 12 Post-partum | 117660.87 (33240.095)
  TAF: Second Trimester: number analyzed (Participants) | 14
  TAF: Second Trimester | 62333.17 (37242.307)
  TAF: Third Trimester: number analyzed (Participants) | 16
  TAF: Third Trimester | 53230.98 (16727.325)
  TAF: Week 6 Post-partum: number analyzed (Participants) | 26
  TAF: Week 6 Post-partum | 44440.06 (13678.515)
  TAF: Week 12 Post-partum: number analyzed (Participants) | 30
  TAF: Week 12 Post-partum | 49837.70 (22019.454)

11. Secondary Outcome: PK Parameter: λz of BIC, FTC, and TAF
Description: λz is defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log plasma concentration of drug versus time curve of the drug.
Time Frame: as for outcome 1
Population: Participants in the PK analysis set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
1/h
  BIC: Second Trimester: number analyzed (Participants) | 19
  BIC: Second Trimester | 0.077 (0.0231)
  BIC: Third Trimester: number analyzed (Participants) | 30
  BIC: Third Trimester | 0.068 (0.0125)
  BIC: Week 6 Post-partum: number analyzed (Participants) | 29
  BIC: Week 6 Post-partum | 0.040 (0.0098)
  BIC: Week 12 Post-partum: number analyzed (Participants) | 30
  BIC: Week 12 Post-partum | 0.043 (0.0134)
  FTC: Second Trimester: number analyzed (Participants) | 20
  FTC: Second Trimester | 0.113 (0.0142)
  FTC: Third Trimester: number analyzed (Participants) | 30
  FTC: Third Trimester | 0.112 (0.0173)
  FTC: Week 6 Post-partum: number analyzed (Participants) | 28
  FTC: Week 6 Post-partum | 0.114 (0.0151)
  FTC: Week 12 Post-partum | 0.120 (0.0209)
  TAF: Second Trimester: number analyzed (Participants) | 14
  TAF: Second Trimester | 2.227 (0.7128)
  TAF: Third Trimester: number analyzed (Participants) | 16
  TAF: Third Trimester | 2.550 (0.7519)
  TAF: Week 6 Post-partum: number analyzed (Participants) | 26
  TAF: Week 6 Post-partum | 1.777 (0.4685)
  TAF: Week 12 Post-partum: number analyzed (Participants) | 30
  TAF: Week 12 Post-partum | 1.954 (0.4519)

12. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at the Time of Delivery Using the Missing = Excluded Approach in B/F/TAF Group
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at the time of delivery was analyzed in B/F/TAF group using missing = excluded approach. In this approach, all missing data were excluded in the computation of the percentages (ie, missing data points were excluded from both the numerator and denominator in the computation).
Time Frame: At time of delivery
Population: Full analysis set included all adult participants who enrolled into the study and took at least 1 dose of study drug (B/F/TAF). Participants in the full analysis set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 32
percentage of participants | 100.0 [89.1 to 100.0]

13. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Birth Using the Missing = Excluded Approach in Neonates
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at the time of birth was analyzed in neonates using missing = excluded approach. In this approach, all missing data were excluded in the computation of the percentages (ie, missing data points were excluded from both the numerator and denominator in the computation).
Time Frame: At birth
Population: Neonate full analysis set included neonates who were born to women participating in the study and had been enrolled into the study as well. Participants in the neonate full analysis set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neonates
Number analyzed (Participants) | 2
percentage of participants | 100.0 [15.8 to 100.0]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From birth up to 8 weeks of age for neonates; From enrollment up to 38 weeks + 30 days for B/F/TAF group. Adverse Events: First dose date up to 38 weeks + 30 days for B/F/TAF group
Description: B/F/TAF:Safety analysis set- all adult participants who took at least 1 dose of study drug. Neonates:Safety analysis set- neonates born to women participating & had been enrolled into study. None of neonates participating in study were treated. Adverse events (AE) reported for that group are not treatment emergent (TE). TEAE:any AE with onset on/after start of study drug & no later than 30 days after permanent study drug discontinuation, or any AE leading to premature study drug discontinuation.
Arm/Group | B/F/TAF | Neonates
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29
Serious Adverse Events (participants affected / at risk) | 6/33 | 5/29
Other Adverse Events (participants affected / at risk) | 19/33 | 4/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=33) | Neonates (N=29)
Nonreassuring foetal heart rate pattern (Cardiac disorders) | 1 | 0
Accessory auricle (Congenital, familial and genetic disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Covid-19 (Infections and infestations) | 1 | 0
Sepsis neonatal (Infections and infestations) | 0 | 1
False labour (Pregnancy, puerperium and perinatal conditions) | 3 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=33) | Neonates (N=29)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Foetal heart rate deceleration abnormality (Cardiac disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 4 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT03960645/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT03960645/SAP_001.pdf